CLINICAL TRIAL: NCT01669902
Title: HAQIMONO a Non-interventional National Multicenter Study, Observing RA Patients Treated With Tocilizumab in Mono-therapy, i.e. Without Combination With DMARD
Brief Title: An Observational Study of RoActemra/Actemra (Tocilizumab) in Monotherapy in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28247
Record Dates: First submitted 2012-08-13; First posted 2012-08-21 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter observational study will evaluate the use of RoActemra/Actemra (tocilizumab) in monotherapy in patients with active moderate to severe rheumatoid arthritis unable to use methotrexate. Eligible patients initiated on RoActemra/Actemra treatment will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) ACR criteria
* Patients who for any reason do not take methotrexate and for whom the treating physician has made a decision to prescribe RoActemra/Actemra as monotherapy; patients who commenced RoActemra/Actemra as monotherapy within 8 weeks prior to the enrolment visit may be included
* Concomitant treatment with non-steroidal anti-inflammatory drug (NSAID) or corticosteroids (orally or intra-articularly) is allowed

Exclusion Criteria:

* Patients who have received RoActemra/Actemra more than 8 weeks prior to enrolment visit
* Previous RoActemra/Actemra treatment in a clinical trial or for compassionate use
* Concomitant DMARD treatment for rheumatoid arthritis (e.g. hyroxychloroquine, sulfasalazine, methotrexate, leflunomide, gold compounds, cyclosporine)
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational agent, whichever is longer) before starting RoActemra/Actemra treatment
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active moderate to severe rheumatoid arthritis unable to use methotrexate
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Denmark (6):
  - Esbjerg
  - Holbæk
  - Kolding
  - Køge
  - Svendborg
  - Vejle
- Norway (5):
  - Bergen
  - Gjettum
  - Moss
  - Skien
  - Trondheim
- Sweden (15):
  - Falun
  - Farsta
  - Gothenburg
  - Helsingborg
  - Hudiksvall
  - Jönköping
  - Karlskrona
  - Karlstad
  - Kristianstad
  - Malmo
  - Simrishamn
  - Skövde
  - Trelleborg
  - Uppsala
  - Västerås

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants with rheumatoid arthritis who were considered for or treated with tocilizumab monotherapy within the clinical routine were observed for a period of 6 months.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 107
Completed | 78
Not Completed | 29
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 10
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all data from all participants who received at least one injection with tocilizumab.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Tocilizumab Treatment at Month 6
Time Frame: Month 6
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 107
percentage of participants | 76.6

2. Secondary Outcome: Percentage of Participants With Dose Modifications of Tocilizumab
Description: Dose modification is any change in dose; this also included participants who stopped treatment with tocilizumab.
Time Frame: Baseline to Month 6
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 107
percentage of participants | 36.4

3. Secondary Outcome: Swollen Joint Count (SJC)
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1; total was calculated by adding all the joints for a maximum score of 28. A reduction in number of swollen joints compared to baseline indicates improvement.
Time Frame: Baseline, Month 3, Month 6
Population: The Full Analysis Set (FAS) (swollen joint counts) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for swollen joints. n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Tocilizumab
Number analyzed (Participants) | 83
swollen joint count
  Baseline (n=83) | 5.6 (5.2)
  Month 3 (n=73) | 2.5 (3.1)
  Month 6 (n=63) | 1.8 (2.5)

4. Secondary Outcome: Tender Joint Count (TJC)
Description: Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1; total was calculated by adding all the joints for a maximum score of 28. A reduction in number of tender joints compared to baseline indicates improvement.
Time Frame: Baseline, Month 3, Month 6
Population: The FAS (tender joint counts) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for tender joints. n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Tocilizumab
Number analyzed (Participants) | 83
tender joint count
  Baseline (n=83) | 8.6 (6.9)
  Month 3 (n=73) | 4.5 (5.3)
  Month 6 (n=63) | 3.7 (4.9)

5. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP])
Description: DAS28-4 (CRP) was calculated from the SJC and TJC using the 28 joints count, CRP (milligram per liter [mg/L]) and patient global assessment (PtGA) of disease activity (measured on a 0 to 100 millimeter [mm] Visual Analog Scale [VAS]) where 0=no disease activity and 100=worst disease activity). DAS28-4 (CRP) was calculated using the following formula: DAS28-4 (CRP) = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014*PtGA + 0.96. Total score range: 0 to 10, higher score indicated more disease activity. DAS28-4 (CRP) less than or equal to (<= 3.2) implied low disease activity and greater than (>) 3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (CRP) less than (<) 2.6 = clinical remission.
Time Frame: Baseline, Month 3, Month 6
Population: The FAS (DAS28-4 [CRP]) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for DAS28-4 [CRP] assessment. n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 83
Units on a scale
  Baseline (n=83) | 4.76 (1.31)
  Month 3 (n=69) | 3.17 (1.34)
  Month 6 (n=60) | 2.98 (1.21)

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Based on DAS28-4 (CRP)
Description: DAS28-4 (CRP) was calculated from the SJC and TJC using the 28 joints count, CRP (mg/L) and PtGA of disease activity (measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity). DAS28-4 (CRP) was calculated using the following formula: DAS28-4 (CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014*PtGA + 0.96. Total score range: 0 to 10, higher score indicated more disease activity. DAS28-4 (CRP) <= 3.2 implied low disease activity and > 3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (CRP) < 2.6 = clinical remission.
Time Frame: Month 3 and Month 6
Population: FAS (DAS28-4 [CRP]). N (number of participants analyzed) = participants evaluable for this measure. n = participants evaluable for this measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 69
percentage of participants
  Month 3 (n=69): Clinical remission | 36.2
  Month 6 (n=60): Clinical remission | 40.0

7. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (millimeter per hour [mm/hour]), and PtGA of disease activity (measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity). DAS28-4 (ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*ln(ESR) + 0.014*PtGA. Total score range: 0-10, higher score=more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = clinical remission.
Time Frame: Baseline, Month 3, Month 6
Population: The FAS (DAS28-4 [ESR]) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for DAS28-4 [ESR] assessment. n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 59
Units on a scale
  Baseline (n=59) | 5.03 (1.39)
  Month 3 (n=49) | 2.98 (1.41)
  Month 6 (n=45) | 2.64 (1.34)

8. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Based on DAS28-4 (ESR)
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hour), and PtGA of disease activity (measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity). DAS28-4 (ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*ln(ESR) + 0.014*PtGA. Total score range: 0-10, higher score=more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = clinical remission.
Time Frame: Month 3 and Month 6
Population: FAS (DAS28-4 [ESR]). N (number of participants analyzed) = participants evaluable for this measure. n = participants evaluable for this measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
percentage of participants
  Month 3 (n=49): Clinical remission | 38.8
  Month 6 (n=45) : Clinical remission | 57.8

9. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28-4 (CRP)
Description: The DAS28-4 (CRP) [described in Outcome Measure 5] based EULAR response criteria were used to measure individual response as good, moderate, or no response depending on the extent of change from baseline in DAS28 score and the level of disease activity (low, moderate or high) reached. Good responders: change from baseline >1.2 with DAS28 <= 3.2; moderate responders: change from baseline >1.2 with DAS28 in the range of >3.2 to <=5.1 or change from baseline in the range of >0.6 to <=1.2 with DAS28 in the range of >3.2 to <=5.1 or change from baseline >1.2 with DAS28 >5.1 or change from baseline in the range of >0.6 to <=1.2 with DAS28 <=3.2; non-responders: change from baseline <= 0.6 or change from baseline in the range of >0.6 to <=1.2 with DAS28 >5.1 or change from baseline <=0.6 with DAS28 <=3.2 or in the range of >3.2 to <=5.1.
Time Frame: Month 3 and Month 6
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 69
percentage of participants
  Month 3: Good response (n=69) | 43.5
  Month 3: Moderate response (n=69) | 33.3
  Month 3: No response (n=69) | 23.2
  Month 6: Good response (n=60) | 43.3
  Month 6: Moderate response (n=60) | 33.3
  Month 6: No response (n=60) | 23.3

10. Secondary Outcome: Percentage of Participants With EULAR Response Based on DAS28-4 (ESR)
Description: The DAS28-4 (ESR) [described in Outcome Measure 7] based EULAR response criteria were used to measure individual response as good, moderate, or no response depending on the extent of change from baseline in DAS28 score and the level of disease activity (low, moderate or high) reached. Good responders: change from baseline >1.2 with DAS28 <= 3.2; moderate responders: change from baseline >1.2 with DAS28 in the range of >3.2 to <=5.1 or change from baseline in the range of >0.6 to <=1.2 with DAS28 in the range of >3.2 to <=5.1 or change from baseline >1.2 with DAS28 >5.1 or change from baseline in the range of >0.6 to <=1.2 with DAS28 <=3.2; non-responders: change from baseline <= 0.6 or change from baseline in the range of >0.6 to <=1.2 with DAS28 >5.1 or change from baseline <=0.6 with DAS28 <=3.2 or in the range of >3.2 to <=5.1.
Time Frame: Month 3 and Month 6
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
percentage of participants
  Month 3: Good response (n=49) | 51.0
  Month 3: Moderate response (n=49) | 34.7
  Month 3: No response (n=49) | 14.3
  Month 6: Good response (n=45) | 55.6
  Month 6: Moderate response (n=45) | 31.1
  Month 6: No response (n=45) | 13.3

11. Secondary Outcome: Simplified Disease Activity Index (SDAI)
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and physician global assessment (PGA) assessed on 0-10 centimeter (cm) VAS; 0 = no disease activity and 10 = worst disease activity, and CRP (mg/dL). SDAI total score = 0-86. SDAI <=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity.
Time Frame: Baseline, Month 3, Month 6
Population: The FAS (SDAI) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for SDAI. n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 34
Units on a scale
  Baseline (n=34) | 22.46 (11.33)
  Month 3 (n=31) | 11.48 (9.18)
  Month 6 (n=24) | 10.73 (11.74)

12. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Based on SDAI
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-10 cm VAS; 0 = no disease activity and 10 = worst disease activity, and CRP (mg/dL). SDAI total score = 0-86. SDAI <=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity.
Time Frame: Month 3 and Month 6
Population: FAS (SDAI). N (number of participants analyzed) = participants evaluable for this measure. n = participants evaluable for this measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 31
percentage of participants
  Month 3 (n=31): Clinical remission | 12.9
  Month 6 (n=24): Clinical remission | 16.7

13. Secondary Outcome: Clinical Disease Activity Index (CDAI)
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-10 cm VAS; 0 = no disease activity and 10 = worst disease activity. CDAI total score = 0-76. CDAI <= 2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high (or severe) disease activity.
Time Frame: Baseline, Month 3, Month 6
Population: The FAS (CDAI) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for CDAI. n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 35
Units on a scale
  Baseline (n=35) | 21.3 (10.9)
  Month 3 (n=33) | 10.9 (8.9)
  Month 6 (n=24) | 10.4 (11.1)

14. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Based on CDAI
Description: as for outcome 13
Time Frame: Month 3 and Month 6
Population: FAS (CDAI). N (number of participants analyzed) = participants evaluable for this measure. n = participants evaluable for this measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 33
percentage of participants
  Month 3 (n=33): Clinical remission | 12.1
  Month 3 (n=24): Clinical remission | 16.7

15. Secondary Outcome: Number of Participants With an American College of Rheumatology (ACR) Response
Description: ACR response: improvement in tender or swollen joint counts and improvement in 3 of the following 5 criteria: 1) PGA of disease activity, 2) PtGA of disease activity, 3) patient's assessment of pain, 4) patient's assessment of functional disability via a health assessment questionnaire, and 5) CRP at each visit. ACR response is based on 66/68 total joint count.
Time Frame: Baseline to Month 6
Population: Data for ACR response was not reported because in clinical practice the 66/68 joint evaluation needed for this is not performed in the Sweden, Denmark and Norway, the 28 joint count is performed instead.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

16. Secondary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score
Description: Patient Global Assessment of Disease Activity was measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity.
Time Frame: Baseline, Month 3, Month 6
Population: The FAS (VAS disease activity [patient]) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for VAS disease activity (patient). n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 87
mm
  Baseline (n=87) | 61.6 (21.4)
  Month 3 (n=77) | 41.3 (25.9)
  Month 6 (n=69) | 41.6 (26.3)

17. Secondary Outcome: Physician Global Assessment (PGA) of Disease Activity
Description: Physician Global Assessment of Disease Activity was measured on a 0 to 100 mm VAS where 0=no disease activity and 100=worst disease activity.
Time Frame: Baseline, Month 3, Month 6
Population: The FAS (VAS disease activity [physician] included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for VAS disease activity (physician). n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 42
mm
  Baseline (n=42) | 34.0 (16.4)
  Month 3 (n=37) | 19.1 (17.2)
  Month 6 (n=30) | 15.2 (14.3)

18. Secondary Outcome: Percentage of Participants in a PGA of Disease Activity Score Category
Description: A categorical scale (Lickert scale) with the following categories: none, mild, moderate, severe and maximal was used to evaluate disease activity in clinical practice.
Time Frame: Baseline, Month 3, Month 6
Population: FAS (categorical scale [physician]) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for rheumatoid arthritis illness categorical scale (physician). n = participants evaluable for this measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
percentage of participants
  Baseline: Mild (n=51) | 2.0
  Baseline: Moderate (n=51) | 56.9
  Baseline: Severe (n=51) | 33.3
  Baseline: Maximal (n=51) | 7.8
  Month 3: None (n=46) | 8.7
  Month 3: Mild (n=46) | 52.2
  Month 3: Moderate (n=46) | 28.3
  Month 3: Severe (n=46) | 10.9
  Month 6: None (n=41) | 7.3
  Month 6: Mild (n=46) | 78.0
  Month 6: Moderate (n=46) | 4.9
  Month 6: Severe (n=46) | 9.8

19. Secondary Outcome: Patient Global Assessment of Pain
Description: Patient Global Assessment of Pain was assessed using a 100 mm VAS (0 to 100) where 0 = no pain to 100 = worst possible pain.
Time Frame: Baseline, Month 3, Month 6
Population: The FAS (VAS pain) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for VAS pain. n = participants evaluable for this measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 83
mm
  Baseline (n=83) | 60.5 (22.3)
  Month 3 (n=73) | 38.4 (24.5)
  Month 6 (n=68) | 39.9 (27.1)

20. Secondary Outcome: Percentage of Participants With Morning Stiffness
Description: The percentage of participants with morning stiffness ("yes", "no", or "do not know") was assessed at each visit.
Time Frame: Baseline, Month 3, Month 6
Population: FAS (morning stiffness) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or 6) for morning stiffness. n = participants evaluable for this measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 89
percentage of participants
  Baseline: Yes (n=89) | 55.1
  Baseline: No (n=89) | 9.0
  Baseline: Do Not Know (n=89) | 36.0
  Month 3: Yes (n=80) | 47.5
  Month 3: No (n=80) | 3.8
  Month 3: Do Not Know (n=80) | 48.8
  Month 6: Yes (n=68) | 36.8
  Month 6: No (n=68) | 14.7
  Month 6: Do Not Know (n=68) | 48.5

21. Secondary Outcome: Percentage of Participants With Duration of Morning Stiffness
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness. Duration was recorded as less than (<) 30 minutes, 30 to 60 minutes, 60 to 120 minutes, 120 to 240 minutes, more than (>) 240 minutes, or whole day.
Time Frame: Baseline, Month 3, Month 6
Population: FAS (morning stiffness). N (number of participants analyzed) = participants evaluable for this measure. n = participants evaluable for this measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
percentage of participants
  Baseline: <30 minutes (n=49) | 10.2
  Baseline: 30 to 60 minutes (n=49) | 24.5
  Baseline: 60 to 120 minutes (n=49) | 32.7
  Baseline: 120 to 240 minutes (n=49) | 20.4
  Baseline: >240 minutes (n=49) | 6.1
  Baseline: whole day (n=49) | 6.1
  Month 3: <30 minutes (n=38) | 28.9
  Month 3: 30 to 60 minutes (n=38) | 28.9
  Month 3: 60 to 120 minutes (n=38) | 23.7
  Month 3: 120 to 240 minutes (n=38) | 15.8
  Month 3: >240 minutes (n=38) | 0
  Month 3: whole day (n=38) | 2.6
  Month 6: <30 minutes (n=25) | 44.0
  Month 6: 30 to 60 minutes (n=25) | 28.0
  Month 6: 60 to 120 minutes (n=25) | 4.0
  Month 6: 120 to 240 minutes (n=25) | 20.0
  Month 6: >240 minutes (n=25) | 0
  Month 6: whole day (n=25) | 4.0

22. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Months 3 and 6
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Month 3 and Month 6
Population: The FAS (HAQ) included all data from all participants who had at least a baseline value and one follow up value (Month 3 or Month 6) for HAQ.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 82
units on a scale
  Baseline (n=82) | 1.29 (0.62)
  Change at Month 3 (n=72) | -0.29 (0.53)
  Change at Month 6 (n=58) | -0.21 (0.59)
Statistical Analysis 1: Comparison: Tocilizumab; Change at Month 3; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change at Month 6; Test type: Superiority or Other; p = 0.0357, Wilcoxon signed rank test

23. Secondary Outcome: Percentage of Participants With Concomitant Corticosteroids Treatment
Time Frame: Baseline to Month 6
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 107
percentage of participants | 26.2

24. Secondary Outcome: Number of Participants With Use of Disease-Modifying Anti-Rheumatic Drugs (DMARDs) During the Study
Time Frame: Baseline to Month 6
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 107
participants | 1

ADVERSE EVENTS:
Time Frame: Baseline to Month 6
Description: Safety Analysis Set
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 10/107
Other Adverse Events (participants affected / at risk) | 13/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=107)
Ear infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood lactic acid increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=107)
Nasopharyngitis (Infections and infestations) | 7
Headache (Nervous system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.